CLINICAL TRIAL: NCT00707343
Title: Preliminary Evaluation of the Efficacy of [F-18] Fluorothymidine (FLT) to Differentiate Radiation Necrosis From Tumor Recurrence and as a Marker of Proliferation in Patients With Primary Brain Tumors
Brief Title: [F-18] Fluorothymidine (FLT) Imaging on Patients With Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI20112
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Cancer; Brain Tumors
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Radiation: FLT-PET Imaging

INTERVENTIONS:
Radiation: FLT-PET Imaging — radiopharmaceutical 3'-deoxy-3'-[F-18]fluorothymidine, [F-18]FLT, a radiopharmaceutical that directly assess tumor proliferation using Positron Emission Tomography(PET) in differentiating tumor recurrence from radiation necrosis in a group of patients with glial neoplasms.

SUMMARY:
Despite significant advances in the understanding of brain tumor biology and genetics as well as improvements in surgical techniques, radiotherapy administration, and chemotherapy methods, many primary brain tumors remain incurable. Most primary brain tumors are highly infiltrative neoplasms, and are therefore unlikely to be cured by local treatments such as surgery, focal radiotherapy, radiosurgery or brachytherapy. A particularly problematic aspect of the management of patients with brain tumors is the eventual development of enhancing lesions on MRI after radiation therapy. The treating physician is then left with the dilemma of what this enhancing lesion may represent (radiation necrosis versus recurrent tumor). The differential diagnosis is between recurrent tumor or radiation necrosis however the amount of each contributing to the enhancing mass on MRI is difficult if not impossible to assess. This particular problem is very common and most patients develop some degree of radiation necrosis after therapy with radiation. Differentiation of necrosis from recurrence is particularly challenging. MRI is typically unable to make this important distinction as there is simply an enhancing mass, the etiology of which could be either necrosis or recurrence. Other imaging methods such as FDG-PET have been used but this technique is also complicated in that the normal brain has FDG uptake and it is often difficult to differentiate recurrence from necrosis. [F-18]FLT may prove to be the most reliable method in making this important differentiation (necrosis versus recurrence) as normal brain and necrotic brain do not have proliferative activity and thus no [F-18]FLT uptake whereas tumor will have proliferative activity and thus [F-18]FLT uptake.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the preliminary efficacy of the radiopharmaceutical 3'-deoxy-3'-[F-18]fluorothymidine, [F-18]FLT, a radiopharmaceutical that directly assess tumor proliferation using Positron Emission Tomography (PET) in differentiating tumor recurrence from radiation necrosis in a group of 30 patients with glial neoplasms. This preliminary clinical study will investigate [F-18]FLT in patients with previously treated primary malignant brain tumors (WHO Grade II, III or IV glial-based tumors) who have a new or enlarging enhancing lesion on Gd-MRI and in whom it is not possible to differentiate recurrent tumor from radiation necrosis on the basis of conventional imaging techniques. The ability to make this important differentiation and accurately determine the amount/degree of tumor recurrence from the amount/degree of radiation necrosis in the enhancing mass is critical for the care of treated brain tumor patients and could potentially change patient management once validated as an accurate means of differentiating the amount/degree of radiation necrosis from recurrence.

While the safety of [F-18]FLT has been studied in a many patients to date we will also obtain additional safety data on the use of this agent in patients with primary brain tumors in a cohort of the initial 12 patients to be studied. It is important to emphasize that the potential clinical application of [F-18]FLT imaging in brain tumors must be compared to the current widely used imaging techniques of MRI and PET imaging using the agent, [F-18] fluorodeoxyglucose (FDG).

In this study, [F-18]FLT PET will be used to assess the three goals of this project:

1. Show that imaging with [F-18]FLT and PET will or will not better determine the amount/degree of tumor versus necrosis in the abnormal areas seen on the recent MRI scan and FDG-PET scan.
2. The [F-18]FLT radiopharmaceutical is shown to be safe or not safe in the amount administered in this study.
3. The amount of [F-18]FLT that is seen on the PET study is shown to correlate or not to correlate with other tests used to determine the proliferation of brain tumors in a tissue sample of your newly identified abnormality on MRI in the event that another surgical biopsy or procedure is performed

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (n = 20) with primary brain tumors will be studied.
* All patients will have had previous radiation and may or may not have had chemotherapy for treatment of the primary brain tumor.
* All patients must have either radiological or established histological diagnosis of the following general categories: glioma (grade 2 to grade 4) previously treated with radiation therapy and possibly chemotherapy. It is expected that some of the patients may need a biopsy or neurosurgical procedure for diagnostic and/or therapeutic purposes as necessary treatment of their disease. In those instances the pathologic results will be used for correlation with the imaging findings. Only clinically indicated biopsy and/or surgery will be done and surgery is incidental to inclusion in the protocol.
* Patients must be 18 years or older for inclusion in this study.
* After entry into the study, the initial 12 patients are expected to be followed for at least 1 month after the infusion of [F-18]FLT.
* The patient, if female, must be postmenopausal for a minimum of one year or surgically sterile, or on one of the following methods of birth control for a minimum of one month prior to entry into this study: IUD, oral contraceptives, Depo-Provera or Norplant. These criteria can be waived at the discretion of the investigator if the patient's intracranial tumor is considered life threatening and the one month wait required is not in the best interest of the patient. Negative pregnancy test is accepted.
* Pre-treatment laboratory tests for patients receiving [F-18]FLT must be performed within 14 days prior to study entry. These must no greater or less than 4X the normal upper or lower limits. These will include liver enzymes (SGOT, SGPT, ALK Phos, GGT, LDH), bilirubin (direct and total), amylase, serum electrolytes, CBC with platelets and absolute neutrophil counts, prothrombin time, partial thromboplastin time, BUN, creatinine, and urinalysis.
* Pre-treatment radiological scans/studies (Gd- enhanced MRI and FDG-PET) for patients receiving [F-18]FLT must be performed within 10 days of study entry.

Exclusion Criteria:

* Patients with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible.
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who are pregnant or lactating or who suspect they might be pregnant.
* Adult patients who require monitored anesthesia for PET scanning.
* HIV positive patients due to the previous toxicity noted with FLT in this patient group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-10-31 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Hoffman, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FLT-PET Imaging: [F-18] FLT: All participants enrolled.
  FLT-PET Imaging: radiopharmaceutical 3'-deoxy-3'-[F-18]fluorothymidine, [F-18]FLT, a radiopharmaceutical that directly assess tumor proliferation using Positron Emission Tomography(PET) in differentiating tumor recurrence from radiation necrosis in a group of patients with glial neoplasms.
Period: Overall Study
Arm/Group | FLT-PET Imaging: [F-18] FLT
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FLT-PET Imaging: [F-18] FLT
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 47 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Curve (ROC AUC) Values for PET Imaging Techniques
Description: The ROC AUC represents the probability that tumor recurrence will be differentiated from radiation necrosis.
  Positron Emission Tomography (PET) imaging methods using radiopharmaceutical agents F-18 fluorodeoxyglucose (FDG) and F-18 fluorothymidine (FLT) were used for analysis. For F-18 FDG, the maximum standardized uptake value (SUVmax) with correction for body weight was measured at suspicious area of lesion enhancement. The ratio of F-18 FDG SUVmax of the suspicious lesion to that of the SUVmean of a 1 cm diameter region of normal contralateral white matter was also measured (F-18 FDG ratio lesion: contralateral white matter). For F-18 FLT, the maximum standardized uptake value (SUVmax) was measured at suspicious area of lesion enhancement. Patlak graphical analysis was applied using the metabolite-corrected plasma input function to obtain voxel-wise estimates of the FLT metabolic influx parameter (F-18 FLT Kimax).
Time Frame: 30 minutes for FDG imaging, 70 minutes for FLT imaging acquisition; 2-33 months for lesion outcome confirmation
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | FLT-PET Imaging: [F-18] FLT
Number analyzed (Participants) | 15
Probability
  F-18 FDG ratio lesion: contralateral white matter | 0.98 [0.91 to 1.00]
  F-18 FDG SUVmax | 0.91 [0.75 to 1.00]
  F-18 FLT Kimax | 0.89 [0.69 to 1.00]
  F-18 FLT SUVmax | 0.82 [0.56 to 1.00]

ADVERSE EVENTS:
Arm/Group | FLT-PET Imaging: [F-18] FLT
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes